CLINICAL TRIAL: NCT02827721
Title: Evaluation of Novel Lung Function Parameters in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Dr. Frederik Trinkmann, Principal Investigator, Universitätsmedizin Mannheim
Other Study IDs: MBW-COPD
Record Dates: First submitted 2016-06-30; First posted 2016-07-11 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: COPD; Obstructive Ventilation Disorder; Pulmonary Emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pulmonary Emphysema | interventions — Plethysmography, Whole Body

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- COPD: Patients with known or suspected COPD Patients with known or suspected obstructive ventilation disorder
  Interventions: Device: impulse oscillometry; Device: multiple breath washout test; Device: body plethysmography
- pulmonary healthy controls: Patients without known or suspected pulmonary disease
  Interventions: Device: impulse oscillometry; Device: multiple breath washout test; Device: body plethysmography

INTERVENTIONS:
Device: impulse oscillometry
Device: multiple breath washout test
Device: body plethysmography

SUMMARY:
Current guideline-based criteria defining COPD do not meet the challenges set by the complex pathophysiology of the disease. The investigators therefore aimed to evaluate novel or not widely used diagnostic approaches for the detection and therapeutic monitoring of COPD.

ELIGIBILITY:
Inclusion Criteria:

* known or suspected COPD
* known or suspected obstructive ventilation disorder
* pulmonary healthy controls

Exclusion Criteria:

* pregnancy
* inability to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with indication for routine lung function testing
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-07; Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
lung clearance index (LCI) as determined by multiple breath washout | 30 minutes
airway resistance and reactance (R5, X5, R-D5-20) as determined by impulse oscillometry | 30 minutes

SECONDARY OUTCOMES:
repeatability of lung clearance index (LCI) | 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Mannheim, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No